CLINICAL TRIAL: NCT04691219
Title: Efficacy and Safety of Mulberry Leaves on Glycemic Control in Patients With Obesity and Patients With Type 2 Diabetes
Brief Title: Effects of Mulberry Leaves on Glycemic Control in Patients With Obesity and Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBRTA-Q038h/60
Record Dates: First submitted 2018-03-06; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Mulberry leaves; Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulberry leaves powder plus diet control (Experimental)
  Interventions: Dietary Supplement: Mulberry leaves powder; Behavioral: Diet control
- Diet control alone (Other)
  Interventions: Behavioral: Diet control

INTERVENTIONS:
Dietary Supplement: Mulberry leaves powder — Dried powder of mulberry leaves crude extract containing 12 mg of DNJ will be packed in a sealed packet with light and moisture protection. Participants will be instructed to mix 1 packet of the powder with a half glass (approximately 120 mL) of plain water and ingest thrice daily before meals. Additionally, they will be informed to rinse the glass with more water and drink to ensure that all of the powder will be taken.
  Arms: Mulberry leaves powder plus diet control
Behavioral: Diet control — Participants will be requested for diet control. They will be asked for attending the diet control program, maintaining diet pattern throughout the study period, and recording a 3-day food record. Individual counseling and assessment of compliance will be performed by licensed dietitians every 4 weeks. Diet control is principally based on carbohydrate counting.

SUMMARY:
A 12-week, open-label, randomized, controlled trial investigating effect of mulberry leaves plus lifestyle intervention on glycemic control compare with lifestyle intervention alone in patients with obesity and patients with type 2 diabetes (T2DM)

DETAILED DESCRIPTION:
Diabetes remains a common leading cause of morbidity and mortality among population worldwide over decades. Obesity, a crucial risk factors for developing T2DM, commonly exists with insulin resistance and impaired beta-cell function. Early management in individuals at high risk of T2DM should be therefore considered for preventing or delaying the progression of diabetes and diabetic complications.

Since 1-deoxynojirimycin (DNJ), the major antihyperglycemic compound of mulberry leaves, inhibits alpha-glucosidase activities, ingestion of mulberry leaves results in the suppression of postprandial hyperglycemia. Long-term effects of mulberry leaves on glycemic profiles have been demonstrated in numerous clinical studies; however, the results were controversial. In addition, no study was conducted in patients with obesity. As a result, this open-label, randomized controlled study aims to investigate efficacy and safety of mulberry leaves in combination with lifestyle intervention (diet control) on glycemic control in non-diabetic patients with obesity and patients with early-stage T2DM. Efficacy of the interventions will be assessed based on the changes in glycemic indexes, expression of proteins related to insulin resistance and T2DM, and lipid profiles. Meanwhile, safety will be measured by the changes in renal and hepatic enzymes and patient-self reports. The outcomes will be monitored at 4-week interval throughout 12 weeks of the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Women or men age 20-65 years
2. Have 1 of 3 characteristics as follows;

   * Non-diabetic obese patients (BMI ≥25 kg/m2)
   * Patients with T2DM: drug naïve and newly diagnosed within 6 months before study enrollment
   * Patients with T2DM: inadequate control (A1c ≥7%, but not >8%) with metformin therapy (>1,000 mg/day) alone at least 3 months before study enrollment
3. Well communicate in the Thai language

Exclusion Criteria:

1. Allergy to mulberry leaves products
2. FPG ≥180 mg/dL
3. A1c >8%
4. AST and ALT >40 U/L
5. Cr <0.6 or >1.2 mg/dL
6. BUN >20 mg/dL
7. Existing or having history of gastrointestinal surgery or abnormal conditions affecting digestion and intestinal absorption
8. Existing or having history of hematological disorders, thyroid diseases, CVD, ischemic stroke, CKD, or other uncontrolled and life-threatening conditions
9. Presence of significant diabetic complications
10. Taking drugs, supplements, and herbs affecting blood glucose level: corticosteroids, second-generation antipsychotics, niacin, thiazide diuretics, and ß-blockers, within 1 month before study enrollment
11. Taking unnecessary drugs, supplements, and herbs affecting lipid level within 1 month before study enrollment
12. Women during pregnancy or lactation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-26 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Effect on 2-hour postprandial glucose (PPG) during 75-g oral glucose tolerance test (OGTT) (efficacy) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of the 2-hour PPG (in mg/dL) during 75-g OGTT at week 12
Effect on fasting plasma glucose (FPG) (efficacy) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of FPG (in mg/dL) at week 4, 8, and 12
Effect on glycated hemoglobin (A1C) (efficacy) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of A1C (in %) at week 12

SECONDARY OUTCOMES:
Effect on total cholesterol (efficacy) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of total cholesterol (in mg/dL) at week 12
Effect on high-density lipoprotein cholesterol (HDL-C) (efficacy) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of HDL-C (in mg/dL) at week 12
Effect on triglycerides (efficacy) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of triglycerides (in mg/dL) at week 12
Effect on low-density lipoprotein cholesterol (LDL-C) (efficacy) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of LDL-C (in mg/dL) at week 12
Effect on insulin resistance index (efficacy) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of Homeostasis model assessment indexes of insulin resistance (HOMA-IR) at week 12
Adverse effects on renal function (safety) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of serum creatinine (in mg/dL) at week 12
Adverse effects on hepatic function 1 (safety) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of aspartate aminotransferase (AST) (in units/L) at week 12
Adverse effects on hepatic function 2 (safety) | 12 weeks
  To evaluate difference between the treatment group and the control group, and change from baseline of alanine aminotransferase (ALT) (in units/L) at week 12
Self-reported adverse events (safety) | 12 weeks
  Participants in the treatment group (those who were assigned to administer mulberry leaves) were asked to report adverse events caused by mulberry leaves administration (i.e. constipation, diarrhea, abdominal cramp, bloating, and hypoglycemia) to the researchers.

CONTACTS AND LOCATIONS:
Locations (1):
- Pornanong Aramwit, Bangkok, Thailand